CLINICAL TRIAL: NCT05541549
Title: ASCEND-JC: A Multi-center, Randomized, Double-blind, Phase 2 Study, Evaluating JCPyV-specific T Cell Therapy for the Treatment of PML
Brief Title: A Phase 2 Study Evaluating JCPyV-specific T Cell Therapy for PML
Acronym: ASCEND-JC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cellevolve Bio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210001
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: VST; Virus specific T-Cell; cell therapy; PML; JC virus
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Intervention Model Description: randomized, double- blinded, Phase 2 trial in patients with PML due to JCPyV.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Biological: CE-VST01-JC
- CE-VST01-JC (Experimental)
  Interventions: Biological: CE-VST01-JC

INTERVENTIONS:
Biological: CE-VST01-JC — CE-VST01-JC at a dose of 1 × 10^8 cells administered as an intravenous (IV) infusion every 28 days for 4 total infusions

SUMMARY:
This is a randomized, double-blinded, Phase 2 trial in patients with PML due to JCPyV. Patients will receive treatment with a matched virus-specific T-cell product (CE VST01-JC) or placebo, and will then be monitored for response to therapy.

DETAILED DESCRIPTION:
Progressive multifocal leukoencephalopathy (PML) is a demyelinating disease of the central nervous system caused by JC polyomavirus (JCPyV) occurring in immunocompromised patients who face a disease that is usually progressive and often fatal (Padgett 1971; Tan 2010). Annually, it is estimated that 4,000 people develop PML in the United States and Europe combined (NORD 2015).

This is a randomized, double- blinded, Phase 2 trial in patients with PML due to JCPyV. Patients will receive treatment with a matched virus-specific T-cell product (CE VST01-JC) or placebo, and will then be monitored for response to therapy. The study is designed to evaluate whether CE-VST01-JC infusions will slow and ultimately halt neurological progression in patients with PML compared with placebo as evaluated by modified Rankin Score (mRS).

ELIGIBILITY:
* Male or female subjects aged 18 years or older, with actively progressing PML confirmed by MRI and JCPyV present in CSF or in brain biopsy tissue (diagnosis confirmed according to algorithm diagnostic criteria for PML developed by the American Academy of Neurology).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of CE-VST01-JC on time to disease progression, as measured by mRS (modified Rankin Score) | 1 year

IPD SHARING:
Plan to Share IPD: No